CLINICAL TRIAL: NCT06351618
Title: Swedish Female Ice Hockey Injury Study
Brief Title: Epidemiology of Injuries in the Professional Women's Swedish National IceHockey League Permitted to Body-Checking
Status: Recruiting | Type: Observational
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-06114-01
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Sport Injury; Ice-Skates Accident; Sports Accident; Female Athlete Triad; Female
Keywords: women's health; Ice hockey; Elite sport; Injuries; Bodychecking
MeSH Terms: conditions — Female Athlete Triad Syndrome; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elite female ice hockey players in Sweden
  Interventions: Other: No intervention will be conducted.

INTERVENTIONS:
Other: No intervention will be conducted. — No intervention will be conducted.

SUMMARY:
This research project can contribute to a deeper understanding of injury patterns among professional female ice-hockey players allowed to body check. An understanding of common injury types and mechanisms aids the clinician in diagnosis and management. This information can guide preventative strategies in the areas of education, coaching, rule enforcement, rule modifications, equipment improvement, and sportsmanship. Today, ice hockey is a sport associated with many severe injuries that not only causes suffering and lower quality of life for the athlete, but also costs society a lot of money. Reducing the number and severity of sport-related injuries is therefore of importance. Knowledge of the injury epidemiology of women's hockey could also contribute to better preventive training programs and other injury preventive actions in the sport. Currently, only a minority of all sports medicine research is made on female study participants (26). This research project has the possibility to gain more knowledge about the female athlete, not only applicable for elite hockey-players, but also for female athletes in different disciplines and in youth teams. Knowledge of factors associated with injury could also contribute to better injury preventive actions and highlight subgroups in extra need of future preventive interventions.

ELIGIBILITY:
Inclusion Criteria:

* minimum 16 years of age, registered player in the highest Swedish professional ice hockey league for women, SDHL

Exclusion Criteria:

* age under 16 years.

Ages: 16 Years to 110 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Registered players in SDHL.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Injuries per 1000 training hours | 1 year
Injuries per 1000 game hours | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The Faculty of Medicine at Lund University, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Yes